CLINICAL TRIAL: NCT07171398
Title: Impact of Chronic Ankle Instability on Jumping and Agility Performance in Athletes: A Comparative Cross-Sectional Study
Brief Title: Impact of Chronic Ankle Instability on Jumping and Agility in Athletes
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Manisa Celal Bayar University (Other); Saglik Bilimleri Universitesi (Other); Australian Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: 821c0699143e44f4
Record Dates: First submitted 2025-09-06; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Chronic Ankle Instability; Ankle Sprain; Functional Performance Deficit; Athletic Performance
Keywords: Chronic Ankle Instability (CAI); Lateral Ankle Sprain; Functional Performance Tests; Jumping Ability; Agility; Hop Tests; Countermovement Jump (CMJ); 5-10-5 Agility Test; Deepsport AI Analysis; Volleyball, Basketball, Soccer Athletes
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Ankle Instability (CAI): 16 athletes (9 female, 7 male) with chronic ankle instability. History of ≥1 lateral ankle sprain ≥12 months ago, ≥2 "giving way" episodes in last 6 months, CAIT score ≤24, ≥5 years sport participation (≥3 h/week training).
  Interventions: Other: Functional Performance Testing Battery
- Healthy Control (CG): 16 athletes (3 female, 13 male) without history of ankle sprain or instability. CAIT score ≥25, age/sex/sport matched to CAI group, ≥5 years sport participation (≥3 h/week training).
  Interventions: Other: Functional Performance Testing Battery

INTERVENTIONS:
Other: Functional Performance Testing Battery — Participants performed a standardized battery of sport-specific performance tests during a single laboratory session, including:
  Countermovement Jump (height, power, flight time)
  5-10-5 Pro-Agility Shuttle Test
  Acceleration-Deceleration-Acceleration (ADA) Test
  Side Jump Test
  6-Meter Timed Hop Test
  Single-Leg Hop Test
  Triple Crossover Hop Test
  Lateral Hop Test Performance was assessed using the Deepsport AI program and standard timing/distance protocols. Results compared between CAI and control cohorts.

SUMMARY:
This study investigated how chronic ankle instability (CAI) affects functional performance in athletes compared with healthy controls. CAI is a condition that develops after repeated ankle sprains, leading to ongoing "giving way" episodes, pain, and reduced stability.

A total of 32 athletes participated: 16 with CAI and 16 healthy, age- and sport-matched controls. Participants performed a series of sport-specific functional performance tests, including single-leg hop tests, triple crossover hop, lateral hop, 6-meter timed hop, side jump, countermovement jump (CMJ), the 5-10-5 agility test, and the acceleration-deceleration-acceleration (ADA) test. The Deepsport AI program was used for precise measurement of jumping and agility parameters.

Results showed that athletes with CAI had significantly lower jump height and power, reduced hop distances, and slower times in agility and hopping tests compared to controls. These findings suggest that CAI negatively impacts performance in explosive and multidirectional movements, which are essential in sports such as basketball, volleyball, and soccer. No strong correlation was found between CAIT (Cumberland Ankle Instability Tool) scores and objective performance outcomes, suggesting that subjective reports alone may not fully capture functional deficits.

This study highlights the importance of using both subjective questionnaires and objective tests to evaluate ankle instability in athletes. It also supports the need for rehabilitation programs that include not only balance and proprioception training but also specific exercises to improve jumping, agility, and multidirectional performance.

DETAILED DESCRIPTION:
Chronic ankle instability (CAI) is a frequent consequence of lateral ankle sprains, affecting up to 74% of athletes with previous ankle injuries. It is characterized by recurrent sprains, repeated "giving way" episodes, reduced function, and impaired performance. While CAI has been extensively studied in relation to balance and proprioception, its direct effects on sport-specific performance metrics such as jumping and agility remain less clear.

In this cross-sectional case-control study, 32 athletes were enrolled: 16 athletes with CAI and 16 matched healthy athletes with no history of ankle instability. The CAI group was diagnosed using International Ankle Consortium (IAC) criteria (history of ≥1 lateral ankle sprain ≥12 months prior, ≥2 giving way episodes in the past 6 months, CAIT score ≤24, ≥5 years of sports participation). Controls had CAIT scores ≥25 and no ankle injury history.

The testing battery included:

Hop tests: single-leg hop, 6-meter timed hop, triple crossover hop, and lateral hop.

Agility tests: 5-10-5 pro-agility shuttle and acceleration-deceleration-acceleration (ADA) test.

Jump tests: countermovement jump (height, flight time, power) and side jump test.

Measurements were supported by the Deepsport AI program for objective performance analysis.

ELIGIBILITY:
Inclusion Criteria:

* CAI Group:
* History of at least one significant lateral ankle sprain ≥12 months prior to testing
* At least 2 episodes of ankle "giving way" in the past 6 months
* Cumberland Ankle Instability Tool (CAIT) score ≤24
* Minimum of 5 years of sports participation and ≥3 hours of training per week

Inclusion Criteria - Control Group:

* No history of ankle sprain or ankle instability
* CAIT score ≥25
* Matched to CAI group by age, sex, and sport participation
* Minimum of 5 years of sports participation and ≥3 hours of training per week

Exclusion Criteria:

* History of fracture, surgery, or major injury in the lower extremity within the past year
* Musculoskeletal injury in the knee, hip, or back in the past 3 months
* Neurological or vestibular disorders affecting balance or movement
* Acute ankle pain, swelling, or inflammation at time of testing
* Current use of orthotics or ankle braces during performance testing
* Systemic or cardiovascular disease preventing safe participation

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty-two athletes (16 with chronic ankle instability, 16 healthy controls) aged 18-30 years, recruited from volleyball, basketball, and soccer teams. Participants were matched for training background and sport exposure, with both groups averaging ≥5 years of training history and ≥3 hours of weekly participation.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Countermovement Jump - Jump Height | Single laboratory session (~60 minutes)
  Jump height (cm) measured during countermovement jump using Deepsport AI. Best of 3 trials recorded.
Countermovement Jump - Flight Time | Single laboratory session
  Flight time (s) measured during countermovement jump with Deepsport AI. Best of 3 trials recorded.
Countermovement Jump - Power Output | Single laboratory session
  Power output (W) calculated from CMJ using Deepsport AI (jump force-time algorithm). Best of 3 trials recorded.
5-10-5 Pro-Agility Shuttle - Completion Time | Single session
  Total completion time (s) for the 5-10-5 shuttle test, measured with electronic timing gates. Best of 2 trials recorded.
Acceleration-Deceleration-Acceleration (ADA) - Total Time | Single session
  Total sprint time (s) across 10 m acceleration, 5 m deceleration, and 10 m re-acceleration, measured with Deepsport AI.
Side Jump Test - Completion Time | Single session
  Time (s) to complete 10 consecutive lateral single-leg jumps across a line. Best attempt recorded.
6-Meter Timed Hop - Completion Time | Single session
  Time (s) to hop forward 6 meters on one leg, measured with stopwatch. Best of 3 trials recorded.
Single-Leg Hop - Completion Time | Single session
  Time (s) to hop forward 6 meters on one leg. Best of 3 attempts recorded.
Triple Crossover Hop - Distance | Single session
  Distance (m) covered in 3 consecutive crossover hops over a 15 cm line. Best of 3 trials recorded.
Lateral Hop Test - Distance | Single session
  Distance (m) covered in 3 consecutive lateral hops on one leg. Best of 3 attempts recorded.

OTHER OUTCOMES:
Cumberland Ankle Instability Tool (CAIT) Score | Baseline assessment (same day as testing)
  Self-reported ankle instability using CAIT questionnaire (0-30 points). Lower scores = greater instability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study, including raw test results (jumping, agility, hop test outcomes), CAIT questionnaire scores, and baseline demographic data (age, sex, sport background), will be shared upon reasonable request for academic research purposes.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD and supporting documents will be available beginning 6 months after publication of the trial results. Data will remain available for 5 years following publication.
Access Criteria: Qualified academic researchers may request access to the de-identified dataset, study protocol, and SAP. Requests should be submitted to the corresponding author and will be reviewed by the research team. Access will be granted for scientifically valid proposals and shared via secure data transfer in accordance with institutional and ethical regulations.
URL: https://orcid.org/0000-0002-1524-6295